CLINICAL TRIAL: NCT00231686
Title: Effects of a 6-Months Physical Conditioning Program on Health Status and Physical Activity in Youths and Young Adults With Cystic Fibrosis - MUKOTRAIN
Brief Title: Effects of a 6-Months Physical Conditioning Program in Patients With Cystic Fibrosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Julius-Maximilians University (Other)
Collaborators: Mukoviszidose eV (German CF society) (Unknown); Schweizer CF-Gesellschaft (Swiss CF society) (Unknown); Hannover Medical School (Other); Goethe University (Other); Triemli Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUKOTRAIN
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2005-10-04 (Estimated); Status verified 2005-09

CONDITIONS: Cystic Fibrosis
Keywords: Lung function test; Physical conditioning, human; Physical fitness; Quality of life
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

INTERVENTIONS:
Behavioral: Supervised aerobic training
Behavioral: Supervised strength training
Behavioral: Unsupervised training

SUMMARY:
The purpose of this randomized, controlled trial was to determine whether a (and if so which) physical conditioning program is effective to improve health status, physical activity, and quality of life in patients with cystic fibrosis. A positive effect of physical conditioning was expected.

DETAILED DESCRIPTION:
A high level of physical activity might be beneficial for patients with cystic fibrosis (CF). Several studies have indicated that physical training might improve fitness and lung functions (or, at least, slow the decline in lung functions). However, there are no long-term studies comparing the effects among aerobic training, strength training and no training. Furthermore, motivation to continue a training with little variations between sessions has been shown to decline rapidly. Thus, adherence with such a program may be low. Finally, not all patients feel happy with the same program. Therefore, a home-based individualized sports program might be best suitable to achieve long term benefits. The MUKOTRAIN study is a multicenter randomized controlled trial to determine the effects of a home-based physical training in patients with CF.

Comparisons:

Study A) Patients training aerobically 3 * 30 min per week (supervised in a sports club near their homes) in addition to their baseline physical activity compared to patients training upper and lower body strength 3 * 30 min per week (supervised in a sports club near their homes) compared to patients maintaining their physical activity. The supervised intervention lasted 6 months, thereafter patients were followed for an additional 18 months.

Study B) Patients asked to participate in sport activities at least 3 * 60 min per week (free choice of activities) in addition to their baseline physical activity compared with patients asked to maintain their baseline physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of cystic fibrosis
* Able to engage in intense physical activities

Exclusion Criteria:

* FEV1 <35%predicted
* Esophageal varicosis
* Pulmonary bullae
* Drop in arterial oxygen saturation with exercise <80%
* Non-CF related chronic diseases
* Signs of pulmonary hypertension (ECG and echocardiogram)

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80
Dates: Start 2000-11; Study Completion 2003-05

PRIMARY OUTCOMES:
Change in lung functions determined at 0,3,6,12,18,24 months
Change in exercise capacity determined at 0,3,6,12,18,24
months
Change in physical activity determined at 0,3,6,12,18,24 months
Change in quality of life determined at 0,3,6,12,18,24 months

SECONDARY OUTCOMES:
Change in body fatness at 0,3,6,12,18,24 months

CONTACTS AND LOCATIONS:
Overall Officials: Helge U Hebestreit, MD, Principal Investigator — Julius-Maximilians University, Würzburg, Germany; Susi Kriemler, MD, Principal Investigator — Stadtspital Triemli, Zürich Switzerland
Locations (4):
- Germany (3):
  - Johann Wolfgang Goethe Universität, Frankfurt
  - Medizinische Hochschule, Hanover
  - Children´s Hospital, Julius Maximilians University, Würzburg
- Stadtspital Triemli, Zurich, Switzerland

REFERENCES:
- [Derived] Hebestreit H, Schmid K, Kieser S, Junge S, Ballmann M, Roth K, Hebestreit A, Schenk T, Schindler C, Posselt HG, Kriemler S. Quality of life is associated with physical activity and fitness in cystic fibrosis. BMC Pulm Med. 2014 Feb 27;14:26. doi: 10.1186/1471-2466-14-26. PMID 24571729
- [Derived] Kriemler S, Kieser S, Junge S, Ballmann M, Hebestreit A, Schindler C, Stussi C, Hebestreit H. Effect of supervised training on FEV1 in cystic fibrosis: a randomised controlled trial. J Cyst Fibros. 2013 Dec;12(6):714-20. doi: 10.1016/j.jcf.2013.03.003. Epub 2013 Apr 13. PMID 23588193
- [Derived] Hebestreit H, Kieser S, Junge S, Ballmann M, Hebestreit A, Schindler C, Schenk T, Posselt HG, Kriemler S. Long-term effects of a partially supervised conditioning programme in cystic fibrosis. Eur Respir J. 2010 Mar;35(3):578-83. doi: 10.1183/09031936.00062409. Epub 2009 Jul 30. PMID 19643946